CLINICAL TRIAL: NCT05104463
Title: A Phase 2a, Randomized, Placebo-Controlled, Double-Blind, Crossover Study to Evaluate the Safety, Tolerability and Effects of CST-2032 and CST-107 on Cognition in Subjects With Mild Cognitive Impairment or Mild Dementia Due to Parkinson's or Alzheimer's Disease
Brief Title: A Study of CST-2032 and CST-107 in Subjects With Mild Cognitive Impairment or Mild Dementia Due to Parkinson's or Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CuraSen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CST2032/CST107-CLIN-015
Record Dates: First submitted 2021-10-20; First posted 2021-11-03 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CST-2032 (3mg)/CST-107 (3mg) to Placebo (Experimental): Participants will receive daily doses of CST-2032 (3mg) co-administered with CST-107 (3mg) for 14 days, followed by a washout period of no drug for 7 days, followed by matching placebo for CST-2032 and matching placebo for CST-107 for 14 days.
  Interventions: Drug: CST-2032, matching placebo for CST-2032, CST-107, matching placebo for CST-107
- Placebo to CST-2032 (3mg)/CST-107 (3mg) (Experimental): Participants will receive matching placebo for CST-2032 and matching placebo for CST-107 for 14 days followed by a washout period of no drug for 7 days, followed by daily doses of CST-2032 (3mg) co-administered with CST-107 (3mg) for 14 days.
  Interventions: Drug: CST-2032, matching placebo for CST-2032, CST-107, matching placebo for CST-107

INTERVENTIONS:
Drug: CST-2032, matching placebo for CST-2032, CST-107, matching placebo for CST-107 — CST-2032 and matching placebo white tablets, CST-107 and matching placebo yellow tablets

SUMMARY:
This is a Phase 2a, randomized, placebo-controlled, double-blind, crossover study to evaluate the effects CST-2032 administered with CST-107 on cognition in participants with Mild Cognitive Impairment (MCI) or mild dementia.

DETAILED DESCRIPTION:
Approximately 60 participants will be enrolled in a 2 period, 2-way crossover design following study eligibility confirmation during the screening period. During each treatment period, subjects will receive daily doses of CST-2032 administered with CST-107 or matching placebo for 14 days. Each treatment period will be separated by a washout period of at least 7 days and up to 21 days.

All participants will complete clinical, cognitive and pharmacodynamic assessments during each treatment period. PK blood samples will be collected prior to, during and after study medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥ 50 and ≤ 85 years of age at time of informed consent.
* Diagnosis of mild cognitive impairment OR mild dementia due to either: Parkinson's disease associated with REM sleep behavior disorder (RBD+PD) and positive response to the RBD Single-Question Screen (RBD1Q) and without hallucinations; OR Alzheimer's Disease (AD).
* For participants taking medications: stable dose and regimen for at least 30 days (90 days for anti-psychotic medications) prior to Day -1 and the dose must remain unchanged through the End of Study Visit unless required for management of adverse events (AEs).
* Cognitive decline not primarily caused by vascular, traumatic, or medical problems (alternative causes of cognitive decline are ruled out).
* Adequate visual and auditory abilities and motor skills to perform all aspects of the cognitive and functional assessments.
* Has a spouse or caregiver who can accompany the subject at specified study visits (if required based on cognitive function).
* Montreal Cognitive Assessment (MoCA) score ≥ 14 and ≤ 26.
* Unless confirmed to be azoospermic (vasectomized or secondary to medical cause), males must agree to use a male condom from Day -1 until the End of Study visit when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a condom during each episode of penile-vaginal penetration until after the End of Study Visit.
* Females of childbearing potential (i.e., not postmenopausal or surgically sterile) who have a male partner must have a negative serum pregnancy test result and must agree to one of the following from start of Screening through 30 days after the last study medication administration: use a highly effective method of birth control; or monogamous relationship with a male partner of confirmed sterility; or practice complete abstinence.
* Females of non-childbearing potential may be enrolled if it is documented that they are postmenopausal.
* Body weight greater or equal to 50 kg and body mass index (BMI) between 18 and 35 kg/m^2, inclusive at Screening.
* Stable medical conditions for 30 days prior to Screening visit (e.g., controlled hypertension, dyslipidemia).
* Willing to follow the protocol requirements and comply with protocol restrictions.
* Capable of providing informed consent and complying with study procedures.
* Able to speak, understand and read English.

Exclusion Criteria:

* Participants with poorly controlled hypertension despite lifestyle modifications and/or pharmacotherapy.
* Participants with pulmonary disease, including asthma, or evidence of clinically significant moderate or severe pulmonary symptoms.
* Clinical signs indicating syndromes such as corticobasal degeneration, supranuclear gaze palsy, multiple system atrophy, chronic traumatic encephalopathy, signs of frontotemporal dementia, history of stroke, head injury or encephalitis, cerebellar signs, early severe autonomic involvement, or Babinski sign.
* Current evidence of epilepsy, focal brain lesion, head injury with loss of consciousness or meeting DSM-V diagnostic criteria for psychotic disorders, such as schizophrenia or bipolar disorder, or have unstable concomitant psychiatric symptomatology (participants with psychotic disorders may be enrolled if their condition is effectively managed, i.e., must be receiving stable doses of anti-psychotic medications(s) 90 days prior to randomization and must remain on that dose throughout both treatment periods.)
* Evidence of any significant clinical disorder or laboratory finding (e.g., potassium levels below normal range) that renders the participant unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, moderate and severe impairment of hepatic function (as defined by the National Cancer Institute Organ Dysfunction Working Group), cardiovascular, pulmonary, gastrointestinal, endocrine (including thyrotoxicosis, excluding managed hypo and hyperthyroidism), immunologic, dermatologic, neurologic, musculoskeletal, metabolic, renal, or other systemic disease or laboratory abnormality.
* Participants with a history of malignant disease within 5 years, including solid tumors and hematologic malignancies (exceptions: [a] basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured; [b] low-grade adenocarcinoma of the prostate, which are slow growing, and are unlikely to progress or metastasize during the clinical trial).
* Any clinically significant medical condition or disease as determined by medical history, physical examination 12-lead electrocardiogram (ECG) and clinical laboratory assessments conducted that, in the view of the Principal Investigator, will interfere with participation in the study or interpretation of results.
* Clinically significant abnormalities of 12-lead ECG (as determined by a central reader), including QTcF > 440 ms, for males and females, and/or HR < 50 beats per minute, or evidence of bundle branch blocks, as indicated on the Mean ECG Analysis Report during the screening Period.
* A calculated creatinine clearance of ≤60 mL/min according to the Cockcroft-Gault equation.
* Current use of any prohibited prescription medication, over-the-counter medication, or herbal supplements including green tea products during Screening or throughout study, unless approved by both the Investigator and the Sponsor Medical Monitor.
* Prior and/or concurrent treatment with any investigational drug ≤90 days prior to dosing (Day 1), or ≤5 half-lives of the drug (whichever is longer), or current enrollment in any other study treatment or disease study, except for observational studies.
* Prior and/or concurrent treatment with any beta-AR agonists or beta-AR blockers (includes oral meds, IV or inhaled) or any meds that impact adrenergic signaling within the last month prior to Screening. Participants may be on stable doses of serotonin-noradrenaline reuptake inhibitors (SNRIs), or tricyclic antidepressants (TCAs), or any treatment for ADHD including noradrenaline reuptake inhibitors (NRIs), or amphetamines within the last month prior to Screening.
* A history of heart failure, sinus bradycardia, second- or third-degree heart block, hypokalemia, attack of unconsciousness possibly associated with torsades de points or family history of Long QT Syndrome.
* Known or suspected alcohol or substance abuse within the past 12 months and/or positive test for alcohol or drugs of abuse at Screening or Day -1.
* Suicidal ideation with actual intent or plan ("Yes" answer on the C-SSRS ideation items 4 or 5) within 3 months prior to study Screening.
* Positive screening test for human immunodeficiency virus (HIV), hepatitis C antibody (HCV Ab) or current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] at Screening). Subjects with immunity to hepatitis B (defined as negative HbsAg and positive hepatitis B surface antibody [HbsAb]) are eligible to participate in the study.
* Current infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Females who are breastfeeding.
* Any other reason for which the PI considers it is not in the best interest of the participant to undertake the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — CuraSen Therapeutics, Inc.
Locations (15):
- United States (14):
  - CuraSen Investigational Site, Scottsdale, Arizona
  - CuraSen Investigational Site, Lafayette, California
  - CuraSen Investigational Site, Boca Raton, Florida
  - CuraSen Investigational Site, Bradenton, Florida
  - CuraSen Investigational Site, Lady Lake, Florida
  - CuraSen Investigational Site, Miami, Florida
  - CuraSen Investigational Site, New Port Richey, Florida
  - CuraSen Investigational Site, Winter Park, Florida
  - CuraSen Investigational Site, New York, New York
  - CuraSen Investigational Site, Cincinnati, Ohio
  - CuraSen Investigational Site, Houston, Texas
  - CuraSen Investigational Site, Round Rock, Texas
  - CuraSen Investigational Site, Stafford, Texas
  - CuraSen Investigational Site, Salt Lake City, Utah
- CuraSen Investigational Site, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CST-2032 (3mg)/CST-107 (3mg) to Placebo: Subjects will receive daily doses of CST-2032 (3mg) co-administered with CST-107 (3mg) for 14 days, followed by a washout period of no drug for 7-21 days, followed by placebo for 14 days.
- Placebo to CST-2032 (3mg)/CST-107 (3mg): Subjects will receive placebo for 14 days followed by a washout period of no drug for 7-21 days, followed by daily doses of CST-2032 (3mg) co-administered with CST-107 (3mg) for 14 days.
Period: Overall Study
Arm/Group | CST-2032 (3mg)/CST-107 (3mg) to Placebo | Placebo to CST-2032 (3mg)/CST-107 (3mg)
Started | 32 | 32
Completed | 28 | 27
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled in study.
Groups:
- Overall: All participants enrolled in study
Arm/Group | Overall
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 59
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 8
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events
Description: The number of participants experiencing treatment-emergent adverse events after receiving 3mg CST-2032 co-administered with 3mg CST-107 compared to placebo
Time Frame: Change from Baseline after 14 days of treatment
Population: Safety Set - All participants who received at least 1 dose of blinded study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants following treatment with placebo.
- CST-2032 and CST-107: Participants following treatment with CST-2032 and CST-107.
Arm/Group | Placebo | CST-2032 and CST-107
Number analyzed (Participants) | 59 | 59
Participants | 19 | 20

2. Primary Outcome: Vital Signs
Description: Change from Baseline in supine blood pressure (diastolic blood pressure and systolic blood pressure) after CST-2032 co-administered with CST-107 compared to placebo
Time Frame: Change from Baseline after 14 days of treatment respectively (4 hours post dose)
Population: Safety set - all participants who received at least 1 dose of study drug (CSR-2032, CST-107 or placebo). Participants were reported based on the treatment received. It is noted that whilst all the above participants were included in the overall analysis, there were some participants for whom data was not available at individual timepoints and the resulting corrected number of participants analyzed is presented per parameter below.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- PD Participants - Placebo: Participants with Parkinson's disease, following treatment with placebo.
- PD Participants - CST-2032/CST-107: Participants with Parkinson's disease, following treatment with CST-2032/CST-107
- AD Participants - Placebo: Participants with Alzheimer's disease, following treatment with placebo.
- AD Participants - CST-2032/CST-107: Participants with Alzheimer's disease, following treatment with CST-2032/CST-107
- Overall - Placebo: All participants following treatment with placebo.
- Overall - CST-2032/CST-107: All participants following treatment with CST-2032/CST-107
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST-2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
mmHg
  Systolic blood pressure - Supine Change from Baseline at Day 14: number analyzed (Participants) | 26 | 24 | 32 | 30 | 58 | 54
  Systolic blood pressure - Supine Change from Baseline at Day 14 | -1.1 (22.17) | -5.2 (19.24) | 1.3 (11.18) | 0.6 (9.53) | 0.2 (16.88) | -2.0 (14.79)
  Diastolic blood pressure - Supine Change from Baseline at Day 14: number analyzed (Participants) | 26 | 24 | 32 | 30 | 58 | 54
  Diastolic blood pressure - Supine Change from Baseline at Day 14 | -0.6 (14.77) | -1.6 (12.40) | 1.5 (8.21) | 2.4 (7.25) | 0.6 (11.55) | 0.6 (9.98)

3. Primary Outcome: Electrocardiograms (ECGs)
Description: Change from Baseline in QTc interval using the Fredericia (QTcF) corrections after treatment with CST-2032 co-administered with CST107 compared to placebo
Time Frame: Change from Baseline after 14 days of treatment respectively (4 hour post-dose)
Population: Safety set - all participants who received at least 1 dose of study drug (CST-2032, CST-107 or placebo). Participants were reported based on the treatment received.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Overall - CST2032/CST-107: All participants following treatment with CST2032/CST-107
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
msec | 4.402 (8.5028) | 4.532 (11.3533) | 2.771 (12.5605) | 3.411 (14.4734) | 3.515 (10.8381) | 3.909 (13.0718)

4. Secondary Outcome: Change From Baseline in DSST Score
Description: Change from Baseline in Digit Symbol Substitution Test (DSST) after CST-2032 co-administered with CST-107 compared to placebo. Participants are asked to copy simple graphic symbols that are paired to the digits 1-9 within a specified time period. Using a key, the examinee is asked to draw each symbol under its corresponding number. The examinee's score is determined by the number of symbols correctly drawn within a 90-second time limit. Higher scores indicate better performance.
Time Frame: Change from Baseline after 7 and 14 days of treatment respectively.
Population: Full Analysis Set - All randomized participants who took at least 1 dose of blinded study drug (CST-2032 + CST-107 or placebo). Participants were analyzed according to the treatment assigned at randomization. It is noted that whilst all the above participants were included in the overall analysis, there were some participants for whom data was not available at individual timepoints and the resulting corrected number of participants analyzed is presented per parameter below.
Measure: Least Squares Mean (Standard Error); unit: correct symbols
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST-2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
correct symbols
  Change from Baseline at Day 7: number analyzed (Participants) | 26 | 25 | 32 | 32 | 58 | 56
  Change from Baseline at Day 7 | 2.09 (0.938) | 3.21 (0.949) | 3.07 (0.905) | 3.71 (0.915) | 2.64 (0.669) | 3.45 (0.676)
  Change from Baseline at Day 14: number analyzed (Participants) | 26 | 25 | 32 | 31 | 58 | 59
  Change from Baseline at Day 14 | 2.79 (0.938) | 2.57 (0.949) | 2.95 (0.906) | 4.71 (0.915) | 2.88 (0.669) | 3.71 (0.676)

5. Secondary Outcome: Change From Baseline in DSST Total Incorrect
Description: Change from Baseline in Digit Symbol Substitution Test (DSST) after CST-2032 co-administered with CST-107 compared to placebo. Participants are asked to copy simple graphic symbols that are paired to the digits 1-9 within a specified time period. Using a key, the examinee is asked to draw each symbol under its corresponding number. The incorrect score is the number of symbols incorrectly drawn within a 90-second time limit. Lower scores indicate better performance; negative scores indicate better performance relative to baseline.
Time Frame: Change from Baseline after 7 and 14 days of treatment respectively.
Population: Full Analysis Set - All randomized participants who took at least 1 dose of blinded study drug (CST-2032 + CST-107 or placebo). Partcipants were analyzed according to the treatment assigned at randomization.
Measure: Least Squares Mean (Standard Error); unit: incorrect symbols
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST-2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
incorrect symbols
  Change from Baseline at Day 7: number analyzed (Participants) | 26 | 25 | 32 | 31 | 58 | 56
  Change from Baseline at Day 7 | 1.41 (0.534) | -0.03 (0.543) | -0.69 (0.475) | -1.55 (0.482) | 0.28 (0.359) | -0.81 (0.364)
  Change from Baseline at Day 14: number analyzed (Participants) | 26 | 25 | 32 | 31 | 58 | 56
  Change from Baseline at Day 14 | 0.37 (0.534) | 0.29 (0.543) | -0.89 (0.476) | -1.65 (0.482) | -0.30 (0.359) | -0.72 (0.364)

6. Secondary Outcome: Change From Baseline in CANTAB Stop Signal Reaction Time
Description: Measures response inhibition (impulse control). Participants must respond to an arrow stimulus by selecting one of two options, depending on the direction in which the arrow points. If an audio tone is present, subjects must withhold making that response (inhibition). Lower response times indicate better performance.
Time Frame: Change from Baseline after 7 and 14 days of treatment respectively.
Population: Full Analysis Set - All randomized participants who took at least 1 dose of blinded study drug (CST-2032 + CST-107 or placebo). Participants were analyzed according to the treatment assigned at randomization.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
milliseconds
  Change from Baseline at Day 7: number analyzed (Participants) | 26 | 24 | 32 | 31 | 58 | 55
  Change from Baseline at Day 7 | 30.81 (14.450) | 0.33 (14.975) | -22.27 (14.824) | -12.02 (15.038) | 1.89 (10.521) | -6.39 (10.756)
  Change from Baseline at Day 14: number analyzed (Participants) | 26 | 25 | 32 | 30 | 58 | 55
  Change from Baseline at Day 14 | 31.65 (14.450) | 2.25 (14.697) | -34.68 (14.838) | -8.61 (15.238) | -4.70 (10.524) | -4.07 (10.756)

7. Secondary Outcome: Change From Baseline in CANTAB 5-Choice Reaction Time
Description: Measures changes in cognition by testing psychomotor speed (selecting a flashing circle on a touch tablet screen as quickly as possible). Lower response times indicate better performance.
Time Frame: Change from Baseline after 7 and 14 days of treatment respectively.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST-2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
milliseconds
  Change from Baseline at Day 7: number analyzed (Participants) | 26 | 25 | 32 | 31 | 58 | 56
  Change from Baseline at Day 7 | 1.56 (16.120) | -5.86 (16.370) | -29.53 (9.762) | -18.59 (9.899) | -14.21 (9.529) | -11.06 (9.657)
  Change from Baseline at Day 14: number analyzed (Participants) | 26 | 25 | 32 | 30 | 58 | 55
  Change from Baseline at Day 14 | 0.38 (16.120) | 15.74 (16.370) | -31.09 (9.770) | -40.83 (10.024) | -15.37 (9.533) | -13.21 (9.719)

8. Secondary Outcome: Change From Baseline in CANTAB Paired Associates Learning Tool - Total Adjusted Errors
Description: Measures changes in cognition by testing attention (remembering the location of an abstract pattern on a touch tablet screen). Lower error scores indicate better performance.
Time Frame: Change from Baseline after 7 and 14 days of treatment respectively.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: incorrect patterns
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
incorrect patterns
  Change from Baseline at Day 7: number analyzed (Participants) | 26 | 25 | 32 | 31 | 58 | 56
  Change from Baseline at Day 7 | -4.46 (2.517) | -4.21 (2.546) | 2.05 (2.495) | 0.81 (2.522) | -1.28 (1.785) | -1.87 (1.804)
  Change from Baseline at Day 14: number analyzed (Participants) | 26 | 25 | 32 | 30 | 58 | 55
  Change from Baseline at Day 14 | -0.11 (2.517) | -4.85 (2.546) | 2.69 (2.498) | 0.65 (2.545) | 1.03 (1.785) | -2.22 (1.813)

9. Secondary Outcome: Change From Baseline in CANTAB Delayed Verbal Recognition
Description: Measures changes in cognition by testing memory (recall of 18 words flashed onto a touch tablet screen). An increase in number of words recognized indicates better performance.
Time Frame: Change from Baseline after 7 and 14 days of treatment respectively.
Population: Full Analysis Set - All randomized participants who took at least 1 dose of blinded study drug (CST-2032 + CST-107 or placebo). Subjects were analyzed according to the treatment assigned at randomization.
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
words
  Change from Baseline at Day 7: number analyzed (Participants) | 26 | 25 | 32 | 31 | 58 | 56
  Change from Baseline at Day 7 | 0.15 (0.628) | 0.11 (0.637) | 1.64 (0.744) | 0.14 (0.754) | 1.02 (0.502) | 0.17 (0.509)
  Change from Baseline at Day 14: number analyzed (Participants) | 25 | 25 | 32 | 30 | 57 | 55
  Change from Baseline at Day 14 | -1.08 (0.637) | 0.47 (0.637) | 0.30 (0.745) | -0.07 (0.762) | -0.25 (0.506) | 0.21 (0.512)

10. Secondary Outcome: Change From Baseline in CANTAB Adaptive Tracking Mean Level of Difficulty Achieved
Description: Measures changes in visual and motor coordination and vigilance. In this task, a small circle (target) continuously moves across the screen in a semi-randomized fashion, so as to minimize the subject's ability to predict the trajectory of the target. The subject is instructed to use his/her finger on the touch screen to move a small dot so that it is consistently within the center of the moving target on the screen. During the test, the speed of the circle is adjusted in response to the subject's ability to keep the dot in the circle, ensuring that the test is adapted to the individual subject. The outcome variable was the mean 'difficulty multiplier', which is a calculation adjustment of the participant's accuracy on target relative to current target speed, averaged over the entire testing session. The difficulty multiplier ranges from 0 to 10. Attainment of a higher difficulty multiplier indicates better performance.
Time Frame: Change from Baseline after 7 and 14 days of treatment respectively.
Population: Full Analysis Set - All randomized participants who took at least 1 dose of blinded study treatment (CST-2032 + CST-107 or placebo). Participants were analyzed according to the treatment assigned at randomization.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032/CST-107 | Overall - Placebo | Overall - CST2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
score on a scale
  Change from Baseline at Day 7: number analyzed (Participants) | 26 | 25 | 32 | 31 | 58 | 56
  Change from Baseline at Day 7 | 0.07 (0.091) | 0.11 (0.093) | 0.37 (0.106) | 0.42 (0.106) | 0.22 (0.073) | 0.27 (0.074)
  Change from Baseline at day 14: number analyzed (Participants) | 26 | 25 | 32 | 30 | 58 | 55
  Change from Baseline at day 14 | 0.06 (0.091) | -0.06 (0.093) | 0.36 (0.106) | 0.34 (0.107) | 0.21 (0.073) | 0.15 (0.074)

11. Secondary Outcome: Change From Baseline in Negative Emotional Bias in the Facial Expression Recognition Task (FERT)
Description: Faces with six different basic emotions (happiness, fear, anger, disgust, sadness, surprise) are briefly displayed on a screen and participants are required to indicate the expression of the face via a button-press. Lower response times indicate better performance; negative response times indicate improvement from baseline
Time Frame: Change from Baseline after 14 days of treatment.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Groups:
- AD Participants - Placebo: Participants with Alzheimer's disease following treatment with placebo.
- AD Participants - CST-2032 + CST-107: Participants with Alzheimer's disease following treatment with CST-2032+CST-107.
Arm/Group | PD Participants - Placebo | PD Participants - CST-2032/CST-107 | AD Participants - Placebo | AD Participants - CST-2032 + CST-107 | Overall - Placebo | Overall - CST-2032/CST-107
Number analyzed (Participants) | 26 | 27 | 33 | 32 | 59 | 59
milliseconds
  Reaction Time for Happy Expressions - Change from Baseline at Day 14: number analyzed (Participants) | 25 | 25 | 31 | 30 | 56 | 55
  Reaction Time for Happy Expressions - Change from Baseline at Day 14 | -178.52 (69.13) | -209.77 (68.80) | 23.34 (68.28) | -89.75 (68.97) | -74.41 (44.21) | -145.62 (44.40)
  Reaction Time for Surprise Expressions - Change from Baseline at Day 14: number analyzed (Participants) | 25 | 25 | 31 | 30 | 56 | 55
  Reaction Time for Surprise Expressions - Change from Baseline at Day 14 | -235.05 (85.92) | -186.53 (85.89) | 16.26 (64.96) | -153.09 (65.64) | -96.45 (50.70) | -169.06 (50.99)
  Reaction Time for Negative Expressions - Change from Baseline at Day 14: number analyzed (Participants) | 25 | 25 | 31 | 30 | 56 | 55
  Reaction Time for Negative Expressions - Change from Baseline at Day 14 | -251.85 (66.35) | -222.02 (66.35) | -51.17 (43.41) | -76.53 (43.86) | -135.72 (37.38) | -149.30 (37.42)

ADVERSE EVENTS:
Time Frame: From Day -1 to end of study (up to 48 days).
Arm/Group | Placebo | CST-2032 and CST-107
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 1/59
Other Adverse Events (participants affected / at risk) | 19/59 | 20/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | CST-2032 and CST-107 (N=59)
cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | CST-2032 and CST-107 (N=59)
Lipase increased (Investigations) | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Amylase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Glucose urine (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Protein urine (Investigations) | 1 | 0
Red blood cell count increased (Investigations) | 1 | 0
Urine leukocyte esterase positive (Investigations) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Bowel movement irregularity (Investigations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Covid-19 (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 2
Bradykinesia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 1
Tremor (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Feeling abnormal (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrilation (Cardiac disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Middle insomnia (Psychiatric disorders) | 1 | 0
Rapid eye movement sleep behaviour (Psychiatric disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Central nervous system stimulation (Surgical and medical procedures) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Benign neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT05104463/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT05104463/SAP_001.pdf